CLINICAL TRIAL: NCT06434623
Title: A Multicenter Federal Learning Algorithm to Build an Intelligent Insulin Decision System for Dynamic Glucose Control in Type 2 Diabetic Patients
Brief Title: Federal Learning Algorithm for an Intelligent Insulin Decision System for Dynamic Glucose Control in Type 2 Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20240324025304420
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Medical Records

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients record
  Interventions: Other: patient record

INTERVENTIONS:
Other: patient record — using patient record to construct AI models

SUMMARY:
Constructing an intelligent insulin decision-making system for dynamic glucose control in type 2 diabetes mellitus via a multicentre federated learning algorithm, comparing the performance of the federated learning model, the local model and the initial model, and evaluating their feasibility and safety.

DETAILED DESCRIPTION:
Constructing an intelligent insulin decision-making system for dynamic glucose control in type 2 diabetes mellitus via a multicentre federated learning algorithm, comparing the performance of the federated learning model, the local model and the initial model, and evaluating their feasibility and safety.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes inpatients receiving insulin therapy

Exclusion Criteria:

* use of insulin pumps or glucocorticoids during hospitalisation
* less than two days of insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes who
Sampling Method: Non-Probability Sample
Enrollment: 30100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
the accuracy of AI models | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Professor, Study Director — Fudan University

IPD SHARING:
Plan to Share IPD: Undecided